CLINICAL TRIAL: NCT05993533
Title: Comparison of the 'CTR' Ratio With Standard Haemostasis Parameters in the Follow-up of Patients Undergoing Heparin Therapy
Acronym: QuantiXa
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Direction Centrale du Service de Santé des Armées (Other)
Responsible Party: Sponsor
Other Study IDs: 2022PPRC04; 2023-A00466-39 (Other: IDRCB)
Record Dates: First submitted 2023-08-07; First posted 2023-08-15 (Actual); Last update posted 2023-08-15 (Actual); Status verified 2023-08

CONDITIONS: Venous Thromboembolic Disease
Keywords: Anti Xa activity; heparin treatment

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The Quantra(r) hemostasis analyzer (Stago) is a recent addition to the family of global hemostasis tests. It uses ultrasound-based technology to characterize the viscoelastic properties of a whole blood sample during coagulation. The Qplus(r) cartridge consists of independent channels, each containing different reagents that provide parallel measurements of 6 parameters.

This global test takes into account cellular elements such as platelets and red blood cells in clot formation, and also explores fibrinolysis. In addition, this test is of particular interest in delocalized biology, i.e. at the patient's bedside, and avoids the time-consuming laboratory centrifugation stage required for routine analyzers.

In practice, this test has been developed to monitor haemostasis in patients who may present with a range of coagulopathies of various etiologies, but also in the management of haemorrhagic patients, in order to adapt the administration of blood products in particular.

The Quantra (r) analyzer could therefore be of interest since it could be deployed in overseas operations to manage war casualties.

Recent studies (EACTAIC-ICCVA congress, October 2021) have shown that there is a good correlation between anti-Xa activity and the CTR (coagulation time ratio) parameter of the Quantra cartridge Qplus (TM), suggesting that this automated system could be used to manage anticoagulant therapy.

ELIGIBILITY:
Inclusion Criteria:

* Patients over 18 and affiliated to the french social security system
* Patients on curative heparin (low molecular weight heparin or non-fractionated heparin) for whom anti-Xa activity is prescribed or planned by the clinician
* Samples taken between working hours
* No opposition to study participation

Exclusion Criteria:

* Patients unable to consent
* Anti-Xa activity not prescribed
* Patients on another anticoagulant treatment or not anticoagulated about it
* Samples taken during non-working hours
* Pregnant or breast-feeding women
* Insufficient language level for understanding the information note

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population is composed by hospitalized subjects under heparin therapy and who needs to undergo a blood control
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2023-06-22 (Actual); Primary Completion 2023-12-22 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Correlation between anti-Xa activity and 'CTR' parameter | Through study completion (6 months)
  The primary outcome is to compare anti-Xa activity results with the CTR (coagulation time ratio) parameter of the Qplus(r) cartridge

CONTACTS AND LOCATIONS:
Locations (1):
- HIA Bégin, Saint-Mandé, France